CLINICAL TRIAL: NCT03471429
Title: Canine-assisted ANxiety Reduction IN Emergency
Acronym: CANINE
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: CANINE
Record Dates: First submitted 2018-02-20; First posted 2018-03-20 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-02

CONDITIONS: Anxiety
Keywords: Anxiety; Dog; Canine; Therapy; Depression; Pain
MeSH Terms: conditions — Anxiety Disorders; Depression; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dog: Patient sees therapy dog for 15 minutes, which is standard of care at this hospital.
- No Dog: Patient receives standard of care

SUMMARY:
The purpose of this study is to see if dogs can reduce the anxiety level of patients in the emergency department.

DETAILED DESCRIPTION:
Patients will score their pain, anxiety, and depression. A dog will then come into the patient's room for approximately 15 minutes after which the patient will score his/her pain, anxiety, and depression again.

ELIGIBILITY:
Inclusion Criteria:

* Research staff will screen for inclusion criterion by asking the care providers if they agree with this statement, "I believe this patient is experiencing moderate or greater anxiety".

Exclusion Criteria:

* Extreme intoxication, agitation that precludes conversation with the patient, fear of dogs, dog bite, allergy to dogs.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled from Emergency Department that are 18 or older with moderate or greater anxiety, per physician Gestalt.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Anxiety reduction from Scale | 30 mins
  reduction in anxiety score (0-10). 0=balanced mood (least anxiety) 2= slight fear and worry 4=mild fear and worry 6= moderate worry, physical agitation 8=Feeling really bad, at the edge 10=out of control behavior, self-harm (worst anxiety)

SECONDARY OUTCOMES:
Pain reduction from Wong Baker faces scale | 30 mins
  reduction in pain score (0-10). 0=no hurt (least pain) 2= Hurts little bit 4= Hurts little more 6= Hurts even more 8= Hurts whole lot 10=out of control behavior, self-harm (hurts worst)
Depression reduction from scale | 30 mins
  reduction in depression score (0-10). 0= Balanced mood (least depressed) 2= Slightly depressed 4= Mildly depressed 6= Definite malaise 8= Feeling reall bad, at the edge 10=Despair, suicidal feelings (worst depressed)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kline JA, Fisher MA, Pettit KL, Linville CT, Beck AM. Controlled clinical trial of canine therapy versus usual care to reduce patient anxiety in the emergency department. PLoS One. 2019 Jan 9;14(1):e0209232. doi: 10.1371/journal.pone.0209232. eCollection 2019. PMID 30625184